CLINICAL TRIAL: NCT01462422
Title: Two Community Strategies Comparing Use of Misoprostol for Secondary Prevention to Primary Prevention for Postpartum Hemorrhage: A Randomized Cluster Non-Inferiority Study in Bijapur District, Karnataka, India
Brief Title: Misoprostol for Secondary Prevention of Postpartum Hemorrhage at the Community Level in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Sri B. M. Patil Medical College, Bijapur, Karnataka, India (Unknown); Jawaharlal Nehru Medical College (Other); University of Illinois at Chicago (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2.4.16
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Prevention; Misoprostol; Developing countries; Nurse midwife
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary prevention (Other)
  Interventions: Drug: Misoprostol
- Secondary Prevention (Other)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Selective administration of 800 mcg sublingual misoprostol to women with at least 350 mL blood loss within 1 hour following delivery
  Arms: Secondary Prevention
Drug: Misoprostol — Universal administration of 600 mcg oral misoprostol given to all women within 5 minutes of delivery of the baby
  Arms: Primary prevention

SUMMARY:
This study compares two community-level strategies: selective administration of 800 mcg sublingual misoprostol to women at 350 mL blood loss for secondary prevention of postpartum hemorrhage (PPH) with universal use of 600 mcg oral misoprostol at the time of delivery for primary prevention of PPH. The study hypothesizes that at community-level births, secondary prevention for women is non-inferior (based on clinical parameters) to universal prophylaxis provided to women for primary prevention of PPH. This cluster-design non-inferiority trial has the potential to inform service delivery programs on clinical outcomes, program feasibility, cost and acceptability of two different community models of PPH care using misoprostol.

DETAILED DESCRIPTION:
Rationale for Research: There is an absence of concrete data on the programmatic and cost-effectiveness of different service delivery models for prevention and treatment of postpartum hemorrhage with misoprostol, prompting a discussion of whether resources are best spent on misoprostol for primary prevention at lower levels (with treatment carried out at higher levels via referral) or whether immediate proactive treatment strategies should be considered. As the training and policy implications of universal prevention versus selective treatment approaches vary, simple and effective service delivery models are urgently needed to help governments and organizations decide how to best focus their limited resources. This study proposes to study the efficacy of a hybrid strategy (i.e., secondary prevention) that combines elements of prevention and treatment. Results of this study could provide a new model of care that will medicate fewer women, save costs and address the clinical conundrum of guessing at the safety of administering a prevention dose of misoprostol followed quickly by a larger treatment dose.

Study design: This randomized cluster trial will recruit women with deliveries attended by auxiliary nurse midwives (ANMs) that occur at homes or at health sub-centers. ANMs will be randomized to administer the intervention as described in the primary or secondary prevention arm.

ELIGIBILITY:
Inclusion Criteria:

1. delivering at home or sub-center with an auxilliary nurse midwife (ANM)
2. able and willing to provide informed consent
3. meeting Ministry of Health Guidelines for home or sub-center delivery

Exclusion Criteria:

1. high-risk pregnancy

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3032 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of women with post-delivery hemoglobin ≤ 7.8 gm/dL | 72 hours (plus or minus 8 hours) after delivery
  A 20% rate of post delivery Hb ≤7.8 gm/dL in the study arm with women receiving selective administration of 800 mcg sublingual misoprostol is non-inferior to a 13% rate of post delivery Hb ≤ 7.8 gm/dL in the study arm with women receiving universal 600 mcg oral misoprostol prophylaxis.

SECONDARY OUTCOMES:
Rate of transfer to referral facilities for PPH | within 72 hours (plus or minus 8 hours) after delivery
  Proportion of women who are transferred from the location of delivery to higher level of care because the birth attendent diagnosed or suspected PPH.
Rate of PPH | within 1 hour after delivery
  Proportion of women with 500 mL-999 mL blood loss following delivery, as measured by a calibrated blood collection drape.
Rate of severe PPH | within 1 hour after delivery
  Proportion of women with > 1000 mL blood loss following delivery, as measured by a calibrated blood collection drape.
Rate of adverse events | Within 72 hours (plus or minus 8 hours) after delivery
  Adverse events include prolonged hospitalization, permanent or serious disability, additional threat to life, or death.
Mean blood loss | 1 hour after delivery
  Blood loss will be measured using a blood collection drape, calibrated at 50 mL intervals.
Rate of additional interventions needed to control bleeding | within 72 hours (plus or minus 8 hours) after delivery
  Addtional interventions include administration of other uterotonics (e.g., oxytocin), IV fluids, comprehensive emergency obstetric care, blood transfusion and surgery
Cost-effectiveness | 72 hours (plus or minus 8 hours) after delivery
  The cost-effectiveness of the two interventions will be compared. The cost-effectiveness measure will utilize information collected on cost of the study drug, materials used to control bleeding, and the cost of transfer and subsequent care received by women who are in in need of higher level care.
Proportion of women reporting known side effects of misoprostol | 1 hour after delivery
  Recognized side-effects of misoprostol include: Shivering, fever, headache, nausea, vomiting and diarrhea. Rare side effects include: abdominal pain from uterine cramping, seizures and palpitations (only with overdosing). All women in both study arms, including those in the secondary prevention arm who do not receive the study drug, will be asked if they experienced any of these symptoms.
Acceptability of intervention to women | 72 hours (plus or minus 8 hours) after delivery
  A brief exit interview will be conducted with participants to assess their acceptability of the intervention, including tolerability of any side effects experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Sheila Raghavan, MSc, Principal Investigator — Gynuity Health Projects; Stacie Gellar, PhD, Principal Investigator — University of Illinois at Chicago; Suellen Miller, PhD, CNM, Principal Investigator — University of California, San Francisco; Shivaprasad S Goudar, MD, MHPE, Principal Investigator — Jawaharlal Nehru Medical College
Locations (1):
- Deliveries at health sub-centers and homes, Vijayapura, Karnataka, India

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518
- See also: Gynuity Health Projects website — http://www.gynuity.org